CLINICAL TRIAL: NCT02076139
Title: Pilot Clinical Trial, Double-blind, Randomized, Placebo Controlled and Masked to Evaluate the Tolerability and Immunogenicity of Nyaditum Resae® Probiotic Administered to Adults With or Without Latent Tuberculosis Infection
Brief Title: Safety and Immunogenicity of Nyaditum Resae® Probiotic to Protect From Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manresana de Micobacteriologia, SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NYADATREG
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2017-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; treg; tolerance; probiotic; mycobacteria
MeSH Terms: conditions — Tuberculosis; Mycobacterium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nyaditum resae® 10e4 (Experimental): The subjects will receive 1 drinkable vial (4mL) per day during 14 days. Each vial contains 10e4 Colony-forming units (CFUs) of Nyaditum resae®.
  Interventions: Dietary Supplement: Nyaditum resae® 10e4
- Nyaditum resae® 10e5 (Experimental): The subjects will receive 1 drinkable vial (4mL) per day during 14 days. Each vial contains 10e5 CFUs of Nyaditum resae®.
  Interventions: Dietary Supplement: Nyaditum resae® 10e5
- Placebo (Placebo Comparator): The subjects will receive 1 drinkable vial (4mL) of distilled water per day during 14 days.
  Interventions: Other: Distilled water

INTERVENTIONS:
Dietary Supplement: Nyaditum resae® 10e4
  Arms: Nyaditum resae® 10e4
Dietary Supplement: Nyaditum resae® 10e5
  Arms: Nyaditum resae® 10e5
Other: Distilled water
  Arms: Placebo

SUMMARY:
This is a double-blind, masked, compared with placebo clinical trial in healthy volunteers with or without tuberculosis infection. This trial aims to study the effect of the probiotic Nyaditum resae® at the level of specific Regulatory T cells (Treg) memory cells one week after the first administration and the global tolerability of the treatment. Nyaditum resae® is a preparation in the form of drinkable vials containing heat-killed environmental mycobacteria. The overall objective of the study is the effect of Nyaditum resae® on immunity, which could reduce the risk of developing active tuberculosis.

DETAILED DESCRIPTION:
The incidence of tuberculosis is still a problem of the first magnitude. Every year 1.5 million people die; there are 10 million cases of illness and 100 million new infected. The growing problem of multiresistance is to be added, remaining so prevalent: 700,000 patients, a figure that increases annually with 100,000 people. Prevention of tuberculosis is currently very difficult because it is a disease caused by a bacillus (Mycobacterium tuberculosis) that is transmitted by air: No risk factor for becoming infected has been identified and there is still no prophylactic vaccine that prevents from infection. One of the most characteristic aspects of tuberculosis is that the majority (90-95 %) of people without immunity alterations do not develop the disease after being infected. As for people who do develop the disease, it is still not known why they develop it.

A group of researchers from the Institut Germans Trias i Pujol recently discovered a mechanism that explains this trend. In short, what happens is that certain people create a too strong inflammatory response against tuberculosis bacillus, which ends up creating massive destruction of the tissue that is around the bacillus and brings the characteristic lesion of tuberculosis: tuberculous cavity.

This group of researchers was devising ways to "reeducate" the immune system against the bacillus not make it aggressive. And they did it using two instruments. The first one, an environmental mycobacteria, namely a bacillus of the family of mycobacteria tuberculosis, that usually lives in the water they drink, so that at a greater or lesser extent the investigators already have it in their intestinal flora. The second, inducing a tolerant response, like the investigators do when they eat food. To induce a tolerant response, low and repeated doses of the product make the immune system of the digestive duct "used to" their presence. Thus, when it becomes to find the product, the immune system reacts in a very light and balanced manner, avoiding excessive inflammatory responses. The clearest example is the fact that their immune system "is used" to feed proteins and generates no rejection answers found in the intestinal mucosa.

Hence comes the probiotic Nyaditum resae®, a preparation in the form of drinkable vials, containing a heat-killed environmental mycobacteria and thus can generate a cross-immunity with the tuberculosis bacillus. By giving low and repeated dose to generate a tolerant response, which happens when there is an infection by Mycobacterium tuberculosis, so that a balanced immune response is triggered able to reduce the risk of developing active tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent before starting the selection process.
2. Women and men ≥ 18 years.
3. Availability to meet the requirements of the protocol.

Exclusion Criteria:

1. HIV positive.
2. Known immunodeficiencies.
3. Pregnancy and maternal lactation.
4. Active tuberculosis.
5. Enrollment in another clinical trial.
6. Chronic administration of: methotrexate, azathioprine, cyclophosphamide, oral corticosteroids and other immunosuppressive therapies / immunomodulatory .
7. Administration of blood products or blood derivatives during the 6 months prior to randomization.
8. Detection by the researcher lack of knowledge or willingness to participate and fulfill all the requirements of the protocol.
9. Any other finding that the investigator's opinion, could jeopardize the performance of the protocol or significantly influence the results or interpretation of the effects of probiotic.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Specific Treg memory cells at week 1 | From Baseline to Week 1
  Median increase of specific Treg memory cells at week 1.
Global tolerability of Nyaditum resae ®, proportion of participants with adverse events related to study treatment. | Baseline to week 6
  Proportion of patients presenting adverse events related to study treatment.

SECONDARY OUTCOMES:
Local tolerability (gastrointestinal duct), proportion of participants with gastrointestinal adverse events related to study treatment. | Baseline to week 6
  Proportion of participants presenting gastrointestinal adverse events related to study treatment.
Systemic tolerability (vital signs, physical exam, laboratory tests), proportion of participants with systemic adverse events related to study treatment. | Baseline to week 6
  Proportion of participants presenting systemic adverse events related to study treatment.
Change from Baseline in Specific Treg memory cells at week 2 | From Baseline to Week 2
  Median increase of specific Treg memory cells at week 2.
Change from Baseline in Specific Treg memory cells at month 12 | From Baseline to Month 12
  Median increase of specific Treg memory cells at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Eva Montané, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias I Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Tukvadze N, Cardona P, Vashakidze S, Shubladze N, Avaliani Z, Vilaplana C, Cardona PJ. Development of the food supplement Nyaditum resae as a new tool to reduce the risk of tuberculosis development. Int J Mycobacteriol. 2016 Dec;5 Suppl 1(Suppl 1):S101-S102. doi: 10.1016/j.ijmyco.2016.09.073. Epub 2016 Nov 14. PMID 28043488